CLINICAL TRIAL: NCT00914823
Title: Administration of Kisspeptin to Subjects With Reproductive Disorders
Brief Title: Kisspeptin Administration in the Adult
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, MGH Harvard Center for Reproductive Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2008-P-002486
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Hypogonadotropic Hypogonadism; Kallmann Syndrome; GnRH Deficiency; PCOS; Polycystic Ovarian Syndrome; Hyperprolactinemia
Keywords: reproductive disorders; kisspeptin; hypogonadotropic hypogonadism; Kallmann Syndrome; PCOS
MeSH Terms: conditions — Hypogonadism; Kallmann Syndrome; Polycystic Ovary Syndrome; Hyperprolactinemia | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- kisspeptin, GnRH (Experimental): Intravenous (IV) or subcutaneous (SC) administration of kisspeptin 112-121 and/or administration of GnRH
  Interventions: Drug: kisspeptin 112-121; Drug: GnRH

INTERVENTIONS:
Drug: kisspeptin 112-121 — One or more IV or SC doses of kisspeptin 112-121, and/or short infusion (up to 12 hours) of kisspeptin 112-121
  Other Names: metastin 45-54
Drug: GnRH — One or more IV doses of GnRH, and/or SC administration of GnRH
  Other Names: gonadotropin-releasing hormone

SUMMARY:
The goal of this study is to learn about the role of kisspeptin in the reproductive system. Kisspeptin is a naturally occurring hormone in humans that causes the release of other hormones, including gonadotropin-releasing hormone (GnRH) in the body.

DETAILED DESCRIPTION:
The reproductive hormone GnRH is essential for normal reproductive function. People with idiopathic hypogonadotropic hypogonadism (IHH), hyperprolactinemia, and polycystic ovarian syndrome (PCOS) do not secrete or respond to GnRH in a normal way. In this study, investigators will give participants kisspeptin-a hormone that is naturally found in the human body and is known to be a powerful stimulus of GnRH secretion. They may also give participants GnRH to determine if participants will be able to fully respond to kisspeptin. The goal of this study is to use kisspeptin administration to probe the condition of GnRH neurons in people with various reproductive disorders to better understand the underlying reasons for the disorders. Investigators hope to gain new insights into GnRH neuronal function (or dysfunction) that will lead to better diagnostics in the future.

ELIGIBILITY:
A. Healthy Subjects

All healthy subjects will meet the following criteria:

* normal puberty with respect to onset and pace,
* no chronic diseases,
* no difficulty with blood draws,
* no prescription medications for at least 2 months with the exception of seasonal allergy medications and hormone replacement therapy,
* no illicit drug use or excessive alcohol consumption (< 10 drinks/week),
* no history of a medication reaction requiring emergency medical care,
* normal physical exam and laboratory studies within protocol reference ranges.

Additional criteria based on subject population:

1. Healthy Men:

   * between 21 and 40 years old,
   * normal erectile and ejaculatory function, no history of reproductive disorders,
   * testicular volume >15 ml.
2. Healthy women:

   * between 21 and 40 years old,
   * not breastfeeding or pregnant,
   * menstrual cycles between 25 and 35 days in duration, at least 11 periods/year, with no more than 5 days variability in cycle duration,
   * no evidence for androgen excess (hirsutism or acne),
   * at screening, negative hCG pregnancy test,
   * negative screening for Factor V Leiden for those who might receive estradiol treatment as a part of this study.
3. Healthy postmenopausal women:

   * between 50 and 60 years old,
   * no menstrual periods within the last year,
   * previous history of menstrual cycles between 25 and 35 days in duration, with no more than 5 days variability in cycle duration,
   * if applicable, able to undergo washout from hormone therapy,
   * no evidence for androgen excess (hirsutism or acne),
   * negative screening for Factor V Leiden for those who might receive estradiol treatment as a part of this study.

B. Subjects with Reproductive Disorders

All subjects with reproductive disorders will meet the following criteria:

* 18 years or older,
* all medical conditions stable and well controlled,
* no prescription medications known to affect reproductive endocrine function for at least 2 months except for medications used to treat the subject's reproductive condition,
* no history of a medication reaction requiring emergency medical care,
* no illicit drug use or excessive alcohol consumption (<10 drinks/week),
* for women, not breastfeeding or pregnant,
* if applicable, able to undergo appropriate washout from hormone therapy,
* normal physical exam and laboratory studies within protocol reference ranges,
* for women, at time of screening negative hCG pregnancy test.

Additional criteria based on subject population:

1. Men and women with hypogonadotropic hypogonadism,

   * Confirmed diagnosis by low sex steroids in the setting of low or inappropriately normal gonadotropins,
   * If needed, additional labs and imaging tests may be performed.
2. Women with Polycystic Ovarian Syndrome (PCOS)

   * Confirmed diagnosis of PCOS,
   * If needed, additional labs and imaging tests may be performed.
3. Men and women with hyperprolactinemia

   * confirmed diagnosis of elevated levels of prolactin measured via blood test,
   * no pituitary adenoma OR a microprolactinoma (<10 mm). Patients with a macroprolactinoma confirmed on MRI imaging will be excluded,
   * willing to complete a dopamine agonist washout.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2009-06-23 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Average change in luteinizing hormone (LH) in response to kisspeptin | Within 30 minutes of administration

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie B Seminara, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galbiati F, Plessow F, Plummer L, Campbell MB, Nazarloo S, Carter CS, Davis JM, Miller KK, Carroll RS, Kaiser UB, Seminara SB, Aulinas A, Lawson EA. Intravenous kisspeptin 112-121 bolus does not acutely impact circulating vasopressin in humans. J Neuroendocrinol. 2026 Jan;38(1):e70114. doi: 10.1111/jne.70114. Epub 2025 Nov 22. PMID 41273106
- [Derived] Galbiati F, Plessow F, Plummer L, Campbell MB, Nazarloo S, Carter CS, Carroll RS, Kim HK, Pereira SA, Paulis D, Davis JM, Miller KK, Kaiser UB, Seminara SB, Aulinas A, Lawson EA. Sex-dependent increases in oxytocin levels in response to intravenous kisspeptin in humans. Eur J Endocrinol. 2025 Mar 3;192(3):K24-K29. doi: 10.1093/ejendo/lvaf001. PMID 39965102
- [Derived] Lippincott MF, Leon S, Chan YM, Fergani C, Talbi R, Farooqi IS, Jones CM, Arlt W, Stewart SE, Cole TR, Terasawa E, Hall JE, Shaw ND, Navarro VM, Seminara SB. Hypothalamic Reproductive Endocrine Pulse Generator Activity Independent of Neurokinin B and Dynorphin Signaling. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4304-4318. doi: 10.1210/jc.2019-00146. PMID 31132118
- [Derived] Chan YM, Lippincott MF, Butler JP, Sidhoum VF, Li CX, Plummer L, Seminara SB. Exogenous kisspeptin administration as a probe of GnRH neuronal function in patients with idiopathic hypogonadotropic hypogonadism. J Clin Endocrinol Metab. 2014 Dec;99(12):E2762-71. doi: 10.1210/jc.2014-2233. PMID 25226293